CLINICAL TRIAL: NCT02941419
Title: Safety and Efficacy of Platelet Lysate for Therapeutic Angiogenesis in Patients With Peripheral Arterial Disease
Brief Title: Treatment of PAD by Platelet Lysate for Therapeutic Angiogenesis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Jordan (Other)
Responsible Party: Principal Investigator, Moath AlSmady, Researcher, University of Jordan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PADUJCTC
Record Dates: First submitted 2016-10-19; First posted 2016-10-21 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Critical Limb Ischemia
Keywords: Platelet lysate; Critical limb ischemia; Peripheral arterial disease
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia; Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Platelet lysate injection (Experimental): Injection of platelet lysate intramuscularly in the gastrocnemius muscle
  Interventions: Biological: Platelet lysate

INTERVENTIONS:
Biological: Platelet lysate — Autologous intramuscular platelet lysate injection for patients with peripheral arterial disease

SUMMARY:
Induction of autologous angiogenesis in patients with critical limb ischemia using platelet lysate.

DETAILED DESCRIPTION:
Ten male and female patients diagnosed with Peripheral artery disease (PAD), will be recruited. This diagnosis will be based on medical history, physical examinations, laboratory tests, and specific diagnostic tests. Patients qualified for this study, are patients with distal extremity ischemia indicated by claudication and rest pain present for a minimum of 4 weeks without evidence of improvement in response to conventional drug therapy; showed angiographic evidence of PAD in the affected limb; and were not candidates for surgical revascularization. Platelet lysate will be injected intramuscularly at different sites of the gastrocnemius muscle. The purpose of this study is to evaluate the safety and efficacy of platelet lysate injections into ischematic limbs of patients with PAD.

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to give informed consent, and to be available for all baseline treatment and follow up examinations required by the protocol.
* Gender: Male or female.
* Established Peripheral arterial disease, clinically and hemodynamically confirmed as per Rutherford 3, 4 and
* History of intermittent claudication for > eight weeks.
* Limited exercise due to moderate to severe claudication.
* Resting ankle brachial index (ABI) < 0.85, toe pressure ≤ 60 mm Hg, Toe brachial index (TBI) <0.6, or Trans-cutaneous oxygen pressure (TcPO2) ≤ 60 mmHg in the foot.
* Not eligible for surgical or radiological revascularization.
* In case of diabetic patients, he/she should be on medication and fairly controlled (HbA1c <10%).
* Normal liver enzymes, serum creatinine < 1.4
* Normal platelet count.
* On regular medication for hypertension if any.
* No evidence of malignancy
* Low Questionnaire scores.
* Body mass index <30.

Exclusion Criteria:

* Women with child bearing potential, pregnant and lactating women.
* Rheumatoid Arthritis.
* History of neoplasm or malignancy in the past 10 years.
* Reported unstable cardiovascular disease, heart failure or symptomatic postural hypotension within 6 months before screening.
* Leg edema
* Inflammatory or progressive fibrotic disorder
* Renal insufficiency or failure
* History of infectious disorder.
* Chronic inflammatory disease
* History of stroke or myocardial infarction ( < 3 months).
* Bleeding or clotting disorder, use of oral anticoagulant therapy (heparin, warfarin).
* Lab values for
* Hemoglobin <10 g/dl.
* Platelet count <100,000.
* Prothrombin time/ partial thromboplastin time (PT/PTT)> 3 seconds.
* Alanine aminotrasferase (ALT) and aspartatet aminotrasferase (AST) > 1.5x of the normal lab value.
* Creatinine ≥ 1.4
* Poorly controlled diabetes (HbA1c ≥10)
* Bilirubin > 1.5x of the normal lab value.
* Systemic autoimmune disease.
* Receiving immunosuppressant medications.
* Uncontrolled hypertension or hypotension.
* Abdominal aortic aneurism > 5 cm.
* Active or untreated Tuberculosis.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2013-03-05 (Actual); Primary Completion 2016-09-15 (Actual); Study Completion 2017-02-09 (Actual)

PRIMARY OUTCOMES:
Assessment the safety of platelet lysate injection | 6 months
  Patients will be assessed for any relevant adverse event resulting from the platelet lysate injection

SECONDARY OUTCOMES:
Assessment the efficacy of platelet lysate injection | 6 months
  Assessing the therapeutic benefit of all four platelet lysate injections by ankle brachial index (ABI).

IPD SHARING:
Plan to Share IPD: No